CLINICAL TRIAL: NCT03185728
Title: iLook Out for Child Abuse: An Innovative Learning Module for Childcare Providers
Acronym: iLookOut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: University of Oklahoma (Other); Penn State University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Benjamin H. Levi, Professor, Department of Humanities and Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB-4740; R01HD088448-01 (NIH)
Record Dates: First submitted 2017-04-20; First posted 2017-06-14 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Child Abuse
Keywords: Child Abuse; Mandated Reporting; Online Learning; Child Protection; GAMIFICATION; Early Childhood Education

STUDY DESIGN:
Intervention Model Description: Childcare sites will be randomized to one of 3 study arms, and we will use a stepped wedge design to recruit patients to complete one of two interventions. During the first year of implementation, 1/3 of participants will not be contacted (Control arm). In the other 2 arms, participants will be recruited to complete either the iLookOut intervention or the Standard online mandated reporter training. The next year, participants in the Standard arm will then be asked to complete the iLookOut intervention, and participants in the Control arm will, again, not be incentivized to complete any training. In the final year, participants in the Control arm will be recruited to complete the iLookOut intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iLookOut (Experimental): Online, interactive learning program developed by study team.
  Interventions: Other: iLook Out for Child Abuse
- Standard (Active Comparator): Online mandated reporter training developed by the state of Maine during Y1, then recruited to complete iLookOut during Y2 and Y3.
  Interventions: Other: iLook Out for Child Abuse
- Control (No Intervention): No active recruitment or incentivizing of participants to complete any training on mandated reporting during Y1 and Y2, then recruited to complete iLookOut during Y3.

INTERVENTIONS:
Other: iLook Out for Child Abuse — Online, interactive educational intervention that uses a video-based story-line and "gamification" to teach childcare providers about child abuse and mandated reporting.
  Other Names: iLookOut
  Arms: Standard; iLookOut

SUMMARY:
This five-year study aims to improve childcare provider (CCP) reporting of suspected child abuse by means of an online learning module, iLook Out for Child Abuse. Using an interactive, video-based story-line (along with follow-up activities), iLookOut engages CCPs emotionally and intellectually to take the first step in addressing the epidemic of child abuse -which in the U.S. claims >680,000 confirmed victims annually. The consequences of child abuse can be devastating and long-lasting. The purpose of this study is to establish an evidence-based intervention that can help those who care for young children recognize and report suspected child abuse before irreparable harm occurs.

DETAILED DESCRIPTION:
This 5-year study will evaluate the efficacy of an innovative educational intervention, iLook Out for Child Abuse (iLookOut) for increasing rates of accurate child abuse reporting. Grounded in an Experiential Learning conceptual model, iLookOut is a multi-media, online intervention that engages learners emotionally and intellectually through an interactive, video-based story-line that provides education, challenges learners with decision-points, and gives critical feedback. iLookOut uses "gamification" strategies to promote experiential learning through simulation, problem-solving, and practice opportunities to apply new information and understanding. It also will include follow-up activities that promote retention and integration of new knowledge, as well as help CCPs to remain aware and engaged.

Prior studies have demonstrated that iLookOut significantly improves CCP knowledge and attitudes about reporting suspected child abuse, and is very well received by CCPs. To evaluate its impact on actual reporting behavior, the proposed research will randomize CCP sites in southern Maine (total = ~1,300) to receive iLookOut, Standard training, or Control (no intervention).

The primary goal is to increase the number of CCP reports for which either child abuse is confirmed or social services (e.g., therapeutic services, nutritional assistance) are recommended -as these are the kinds of reports that are likely to actually benefit a child.

The secondary goal is to decrease the proportion of reports that don't offer such benefit, and in particular to decrease costs to the state associated with intake and investigation of non-beneficial reports.

ELIGIBILITY:
Inclusion Criteria:

* Works or volunteers at a childcare facility in Maine (i.e., home-based childcare, childcare center, Head Start facility, nursery school, pre-school)
* 18 years of age or older

Exclusion Criteria:

* Does not work or volunteer at a childcare facility in Maine
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2059 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of "High Quality" reports of suspected child abuse submitted to the State of Maine by childcare providers | 48 months
  Percentage of childcare provider reports (of suspected abuse) to the state of Maine that result in either i) child abuse being confirmed, or ii) social services being recommended for the child/family who was reported.
  We will use Maine's Office of Child and Family Services' criteria for determining what counts as "confirmed child abuse" as well as what counts as a "recommended social service."

SECONDARY OUTCOMES:
Percentage of reports of suspected child abuse submitted to the State of Maine by childcare providers that are "Low Quality" | 48 months
  "Low Quality" reports of suspected abuse are reports to the state of Maine that do not result in either findings of child abuse or recommended social services.
  We will use Maine's Office of Child and Family Services' criteria for determining what counts as "confirmed child abuse" as well as what counts as a "recommended social service."
Financial costs (in U.S. dollars) associated with responding to "Low Quality" reports of suspected abuse that are submitted to the State of Maine by childcare providers | 48 months
  Financial costs (in U.S. dollars) expended by the State of Maine on "Low Quality" reports (submitted by childcare providers during the study period) will be calculated by summing the following:
  i) The average cost to the State of Maine associated with an "Intake call," multiplied by the number of reports of suspected abuse submitted by childcare providers that are screened out (i.e., determined by Intake workers to NOT warrant investigation); and
  ii) The average cost to the State of Maine associated with investigating a report of suspected abuse, multiplied by the number of reports of suspected abuse submitted by childcare providers that are investigated, but NO abuse was confirmed AND no social services were recommended to the child/family that had been reported

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Levi, MD PhD, Study Director — Penn State Milton S. Hershey Medical Center / Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walsh K, Eggins E, Hine L, Mathews B, Kenny MC, Howard S, Ayling N, Dallaston E, Pink E, Vagenas D. Child protection training for professionals to improve reporting of child abuse and neglect. Cochrane Database Syst Rev. 2022 Jul 5;7(7):CD011775. doi: 10.1002/14651858.CD011775.pub2. PMID 35788913

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03185728/Prot_SAP_000.pdf